CLINICAL TRIAL: NCT00714740
Title: Treatment of Patients With the Obstructive Sleep Apnea Syndrome at Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EK-1522
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: apnea, sleep, altitude, hypoxia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea; Hypoxia | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: acetazolamide — acetazolamide 2 times 250mg per day
  Other Names: Diamox

SUMMARY:
The purpose of the study is to investigate the effect of acetazolamide as a treatment for sleep related breathing disturbances in patients with the obstructive sleep apnea syndrome living at low altitude during a sojourn at moderate altitude

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea syndrome, successfully on CPAP therapy
* Residence at low altitude (<800m)
* Obstructive apnea/hypopnea index >20/h and a complaint of excessive daytime sleepiness before introduction of CPAP therapy.
* >15 oxygen desaturations/h (>3% dips) during an ambulatory nocturnal pulse oximetry performed at the end of a 4-night period without CPAP

Exclusion Criteria:

* Sleep disorders other than OSA.
* More than mild cardiovascular disease, unstable or recently diagnosed (within the last 6 months) cardiovascular disease such as arterial hypertension, coronary artery or cerebrovascular disease.
* Any lung disease, pulmonary hypertension.
* Chronic rhinitis.
* Treatment with drugs that affect respiratory center drive (benzodiazepines or other sedatives or sleep inducing drugs, morphine or codeine derivates), stimulants (modafinil, methylphenidate, theophylline)
* Internal, neurologic or psychiatric disease that interfere with sleep quality.
* Previous intolerance to moderate or low altitude (<2600m).
* Exposure to altitudes >1500m for >1 day within the last 4 weeks before the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
sleep disordered breathing, sleep structure, vigilance, subjective sleep quality acute mountain sickness | during treatment while at altitude

SECONDARY OUTCOMES:
blood pressure endothelial function | during treatment while at altitude

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Director — Pulmonary Division, University Hospital Zurich, Switzerland
Locations (1):
- Pulmonary Division, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Nussbaumer-Ochsner Y, Latshang TD, Ulrich S, Kohler M, Thurnheer R, Bloch KE. Patients with obstructive sleep apnea syndrome benefit from acetazolamide during an altitude sojourn: a randomized, placebo-controlled, double-blind trial. Chest. 2012 Jan;141(1):131-138. doi: 10.1378/chest.11-0375. Epub 2011 Jun 9. PMID 21659435
- [Background] Ulrich S, Nussbaumer-Ochsner Y, Vasic I, Hasler E, Latshang TD, Kohler M, Muehlemann T, Wolf M, Bloch KE. Cerebral oxygenation in patients with OSA: effects of hypoxia at altitude and impact of acetazolamide. Chest. 2014 Aug;146(2):299-308. doi: 10.1378/chest.13-2967. PMID 24811331
- [Background] Stadelmann K, Latshang TD, Nussbaumer-Ochsner Y, Tarokh L, Ulrich S, Kohler M, Bloch KE, Achermann P. Impact of acetazolamide and CPAP on cortical activity in obstructive sleep apnea patients. PLoS One. 2014 Apr 7;9(4):e93931. doi: 10.1371/journal.pone.0093931. eCollection 2014. PMID 24710341